CLINICAL TRIAL: NCT01563978
Title: OSKIRA-ABPM: A Multi-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of the Effect of Fostamatinib 100 mg Twice Daily on 24-hour Ambulatory Blood Pressure in Patients With Rheumatoid Arthritis
Brief Title: Study of the Effect of Fostamatinib Twice Daily on Blood Pressure in Patients With Rheumatoid Arthritis
Acronym: Oskira ABPM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4300C00033; 2011-006070-73
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Results first posted 2014-04-14 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dosing Regimen A (Experimental): Oral treatment
  Interventions: Drug: fostamatinib
- Dosing Regimen B (Placebo Comparator): Oral treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fostamatinib — fostamatinib 100 mg twice daily
  Arms: Dosing Regimen A
Drug: placebo — placebo
  Arms: Dosing Regimen B

SUMMARY:
The purpose of this study is to evaluate the effect of fostamatinib compared to placebo on ambulatory blood pressure in patients with active rheumatoid arthritis who are taking a disease-modifying anti-rheumatic drug (DMARD).

The study will last for 57 days.

DETAILED DESCRIPTION:
OSKIRA-ABPM: A Multi-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of the Effect of Fostamatinib 100 mg Twice Daily on 24-hour Ambulatory Blood Pressure in Patients with Rheumatoid Arthritis

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 or over diagnosed with rheumatoid arthritis after the age of 16
* Active rheumatoid arthritis defined as: ≥4 swollen joints and ≥4 tender/painful joints (from 28 joint count) and either erythrocyte sedimentation rate ≥28 mm/h, or C-reactive protein ≥10 mg/L.
* Currently taking one of the following disease-modifying anti-rheumatic drugs: methotrexate, sulfasalazine, hydroxychloroquine or chloroquine.
* Patients without essential hypertension or with essential hypertension if their blood pressure is controlled (<140/90 mmHg) with anti-hypertensive medications being stable at least 4 weeks prior to randomisation.

Exclusion Criteria:

* Females who are pregnant or breastfeeding.
* Certain inflammatory conditions (other than rheumatoid arthritis), connective tissue diseases or chronic pain disorders
* History of liver problems that have required previous investigations
* Evidence of tuberculosis infection
* Conditions that preclude or render difficult the 24-hour ambulatory blood pressure monitoring technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MD PhD, Study Director — AstraZeneca
Locations (56):
- United States (30):
  - Research Site, Huntsville, Alabama
  - Research Site, Huntington Beach, California
  - Research Site, Santa Maria, California
  - Research Site, Trumbull, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Venice, Florida
  - Research Site, Decatur, Georgia
  - Research Site, South Bend, Indiana
  - Research Site, Cumberland, Maryland
  - Research Site, Frederick, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Florissant, Missouri
  - Research Site, Richmond Heights, Missouri
  - Research Site, Freehold, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Lake Oswego, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Nassau Bay, Texas
  - Research Site, Tacoma, Washington
- Bulgaria (2):
  - Research Site, Sevlievo
  - Research Site, Sofia
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hlučín
  - Research Site, Hostivice
  - Research Site, Kladno
  - Research Site, Ostrava-Trebovice
  - Research Site, Prague
- Germany (2):
  - Research Site, Aachen
  - Research Site, Halle
- Poland (8):
  - Research Site, Gdynia
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Kalisz
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Środa Wielkopolska
  - Research Site, Wroclaw
- South Africa (4):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Kempron Park
- Ukraine (4):
  - Research Site, Donetsk
  - Research Site, Kyiv
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 266 patients were enrolled.
Pre-assignment Details: A total of 131 patients failed screening.
Groups:
- FOSTA 100 MG BID: Fostamatinib 100 mg bid, oral treatment
- PLACEBO: Oral treatment
Period: Overall Study
Arm/Group | FOSTA 100 MG BID | PLACEBO
Started | 68 (Patients who received treatment.) | 67 (Patients who received treatment.)
Randomised But Did Not Receive Treatment | 0 | 0
Completed | 64 | 65
Not Completed | 4 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Dev. of study specific discont. criteria | 1 | 0
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOSTA 100 MG BID | PLACEBO | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (12.0) | 54 (13.0) | 54 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 63 | 58 | 121
  Black or African American | 3 | 8 | 11
  Indian or Pakistani | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Mean Ambulatory SBP
Description: ANCOVA=analysis of covariance, BID=twice daily, FAS=full analysis set, IP=investigational product, SBP=systolic blood pressure.
Time Frame: 4 weeks
Population: The FAS includes those randomised patients who received at least 1 dose of IP. Patients were analysed by randomised treatment in accordance with the intention to treat principle.The analysis population for each endpoint includes patients from the FAS still on IP at 4 weeks and with a valid measurement for this type of blood pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 64 | 62
mmHg | 4.3 (7.34) | 1.3 (7.87)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Test type: Superiority or Other; p = 0.023, ANCOVA; Inc. baseline (covariate); treatment, region, prior failure to biologic disease modifying antirheumatic drug & baseline antihypertensive use (factors); Least squares mean treatment difference = 2.93, 95% CI 2-sided [0.40 to 5.45]

2. Secondary Outcome: Change From Baseline in 24-hour Mean Ambulatory DBP
Description: ANCOVA=analysis of covariance, BID=twice daily, DBP=diastolic blood pressure, FAS=full analysis set, IP=investigational product.
Time Frame: 4 weeks
Population: The FAS includes those randomised patients who received at least 1 dose of IP. Patients were analysed by randomised treatment in accordance with the intention to treat principle.The analysis population for each endpoint includes patients from the FAS still on IP at 4 weeks and had a valid measurement for this type of blood pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 64 | 62
mmHg | 4.4 (4.67) | 0.7 (4.41)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean treatment difference = 3.53, 95% CI 2-sided [2.04 to 5.03]

3. Secondary Outcome: Change From Baseline in Mean Daytime and Night-time SBP and DBP by Ambulatory Blood Pressure Monitoring
Description: ANCOVA=analysis of covariance, BID=twice daily, DBP=diastolic blood pressure, FAS=full analysis set, IP=investigational product, SBP=systolic blood pressure.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 64 | 62
mmHg
  Day 28 daytime SBP | 4.9 (8.44) | 1.6 (8.45)
  Day 28 daytime DBP | 4.7 (5.20) | 0.8 (4.89)
  Day 28 night-time SBP | 3.0 (8.59) | 0.9 (9.75)
  Day 28 night-time DBP | 3.7 (6.04) | 0.8 (6.46)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in mean daytime SBP (Day 28); Test type: Superiority or Other; p = 0.020, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 3.30, 95% CI 2-sided [0.53 to 6.08]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in mean daytime DBP (Day 28); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 3.75, 95% CI 2-sided [2.08 to 5.42]
Statistical Analysis 3: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in mean night-time SBP (Day 28); Test type: Superiority or Other; p = 0.179, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 2.07, 95% CI 2-sided [-0.96 to 5.11]
Statistical Analysis 4: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in mean night-time DBP (Day 28); Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 3.14, 95% CI 2-sided [1.13 to 5.14]

4. Secondary Outcome: Change From Baseline in Mean Awake SBP and DBP by Ambulatory Blood Pressure Monitoring
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 63 | 62
mmHg
  Day 28 awake SBP | 4.8 (8.24) | 1.4 (8.37)
  Day 28 awake DBP | 4.8 (4.80) | 0.8 (4.69)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in mean awake SBP (Day 28); Test type: Superiority or Other; p = 0.024, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 3.11, 95% CI 2-sided [0.41 to 5.81]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in mean awake DBP (Day 28); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 3.66, 95% CI 2-sided [2.10 to 5.22]

5. Secondary Outcome: Change From Baseline in Mean Sleeping SBP and DBP by Ambulatory Blood Pressure Monitoring
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 58 | 60
mmHg
  Day 28 sleeping SBP | 2.4 (8.86) | 0.7 (10.12)
  Day 28 sleeping DBP | 2.8 (6.28) | 0.5 (6.72)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in mean sleeping SBP; Test type: Superiority or Other; p = 0.223, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least squares mean treatment difference = 1.99, 95% CI 2-sided [-1.22 to 5.20]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in mean sleeping DBP; Test type: Superiority or Other; p = 0.007, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 2.87, 95% CI 2-sided [0.81 to 4.93]

6. Secondary Outcome: Mean Change From Baseline in Clinic SBP and DBP
Description: Blood pressure was measured in the clinic using an automated blood pressure machine (oscillometric method). Three separate measurements were taken 2 to 5 minutes apart and the mean of the 2nd and 3rd measurements calculated. ANCOVA=analysis of covariance, BID=twice daily, DBP=diastolic blood pressure, FAS=full analysis set, IP=investigational product, SBP=systolic blood pressure.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 64 | 64
mmHg
  Day 29 SBP | 3.8 (11.53) | 2.9 (9.61)
  Day 29 DBP | 2.7 (7.88) | 0.7 (6.72)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in clinic SBP (Day 29); Test type: Superiority or Other; p = 0.200, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 2.24, 95% CI 2-sided [-1.20 to 5.69]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in clinic DBP (Day 29); Test type: Superiority or Other; p = 0.046, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 2.36, 95% CI 2-sided [0.05 to 4.68]

7. Secondary Outcome: Mean Change From Baseline in Morning Pre-dose Home SBP and DBP
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 62 | 59
mmHg
  Weekly average pre-dose SBP (Week 4) | 5.1 (8.53) | -1.3 (6.50)
  Weekly average pre-dose DBP (Week 4) | 4.0 (5.82) | -0.4 (3.78)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in weekly average pre-dose home SBP (Week 4); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 6.31, 95% CI 2-sided [3.60 to 9.03]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in weekly average pre-dose home DBP (Week 4); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 4.58, 95% CI 2-sided [2.91 to 6.25]

8. Secondary Outcome: Mean Change From Baseline in Evening Post-dose Home SBP and DBP
Description: as for outcome 3
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 61 | 59
mmHg
  Weekly average post-dose SBP (Week 4) | 5.3 (9.11) | -1.6 (7.71)
  Weekly average post-dose DBP (Week 4) | 3.7 (5.69) | -1.0 (4.95)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in weekly average post-dose home SBP (Week 4); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 7.22, 95% CI 2-sided [4.29 to 10.16]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID vs PLACEBO; Change from baseline in weekly average post-dose home DBP (Week 4); Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square means treatment difference = 4.74, 95% CI 2-sided [2.90 to 6.59]

9. Secondary Outcome: Mean Change From Completion/Discontinuation to Follow-up in Clinical Measurement of SBP and DBP
Description: BID=twice daily, DBP=diastolic blood pressure, FAS=full analysis set, IP=investigational product, SBP=systolic blood pressure.
Time Frame: Day 29 to Day 36
Population: The FAS includes those randomised patients who received at least 1 dose of IP. Patients were analysed by randomised treatment in accordance with the intention to treat principle. The analysis population for each endpoint includes patients from the FAS still on IP at Day 36 and with a valid measurement for this type of blood pressure assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 64 | 64
mmHg
  SBP | -3.3 (12.32) | -0.5 (9.25)
  DBP | -1.8 (9.56) | -0.6 (6.38)

10. Secondary Outcome: DAS28-CRP Improvement
Description: ANCOVA=analysis of covariance, BID=twice daily, DAS28-CRP=Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (C-reactive protein [CRP]) and the patient's own assessment, FAS=full analysis set, IP=investigational product. Scores can take any positive value with a lower value indicative of a better clinical condition. Mean changes from baseline in DAS28-CRP score are shown at each visit and are presented as decreases from baseline (defined as baseline minus post-baseline) with larger changes indicating a better clinical condition.
Time Frame: 4 weeks
Population: The FAS includes those randomised patients who received at least 1 dose of IP. Patients were analysed by randomised treatment in accordance with the intention to treat principle. The analysis population for each endpoint includes those patients from the FAS who were still on IP at 4 weeks and had a valid measurement for this type of assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID | PLACEBO
Number analyzed (Participants) | 67 | 67
Units on a scale
  Day 8 | 0.8 (0.77) | 0.3 (0.61)
  Day 15 | 1.0 (1.06) | 0.3 (0.77)
  Day 29 | 1.2 (1.06) | 0.5 (1.00)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID vs PLACEBO; Improvement from baseline at Day 29. Non-responder imputation has been applied following premature withdrawal, or any dose of background disease modifying antirheumatic drug increased or any other RA treatment initiated including DMARDs, anti-TNFs or other biologics, or receiving any parenteral steroids, or for patients with no post baseline data; Test type: Superiority or Other; p < 0.001, ANCOVA — Inc. baseline (covariate); treatment, region, prior failure to biologic disease modifying antirheumatic drug & baseline antihypertensive use (factors); Least square means treatment difference = 0.74, 95% CI 2-sided [0.40 to 1.08]

ADVERSE EVENTS:
Arm/Group | FOSTA 100 MG BID | PLACEBO
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67
Other Adverse Events (participants affected / at risk) | 2/68 | 4/67
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID (N=68) | PLACEBO (N=67)
DIARRHOEA (Gastrointestinal disorders) | 2 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review and comment on results communications prior to publication or presentation. Sponsor will be allowed a review period of at least 60 days from submission but can request that the submission be delayed for an additional 90 days from the date of Sponsor's request.